CLINICAL TRIAL: NCT02814669
Title: A Phase Ib, Open-Label Study of the Safety and Tolerability of Atezolizumab in Combination With Radium-223 Dichloride in Patients With Castrate-Resistant Prostate Cancer Who Have Progressed Following Treatment With an Androgen Pathway Inhibitor
Brief Title: Safety and Tolerability of Atezolizumab (ATZ) in Combination With Radium-223 Dichloride (R-223-D) in Metastatic Castrate-Resistant Prostate Cancer (CRPC) Progressed Following Treatment With an Androgen Pathway Inhibitor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO30013; 2015-003606-17 (EudraCT Number)
Record Dates: First submitted 2016-06-20; First posted 2016-06-28 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Castrate-Resistant Prostate Cancer
MeSH Terms: interventions — atezolizumab; radium Ra 223 dichloride

ARMS (6):
- Cohort 1: ATZ + R-223-D (Concurrent) (Experimental): Participants will receive concurrent radium-223 dichloride and atezolizumab for a single-cycle, 28-day dose limiting toxicity (DLT) assessment. If the combination is initially found to be safe and tolerable, additional participants will be randomized to Arms A, B, and C.
  Interventions: Drug: Atezolizumab; Drug: Radium-223 Dichloride
- RT Arm A: ATZ + R-223-D (Concurrent) (Experimental): If Cohort 1 regimen is found to be safe, additional participants will be randomized to this arm (randomized treatment [RT]) to receive concurrent radium-223 dichloride and atezolizumab.
  Interventions: Drug: Atezolizumab; Drug: Radium-223 Dichloride
- RT Arm B: ATZ + R-223-D (Staggered, 28-Day R-223-D Run-In) (Experimental): If Cohort 1 regimen is found to be safe, additional participants will be randomized to this arm to receive radium-223 dichloride in Cycle 1 and radium-223 dichloride and atezolizumab from Cycle 2 onward.
  Interventions: Drug: Atezolizumab; Drug: Radium-223 Dichloride
- RT Arm C: ATZ + R-223-D (Staggered, 28-Day ATZ Run-In) (Experimental): If Cohort 1 regimen is found to be safe, additional participants will be randomized to this arm to receive atezolizumab in Cycle 1 and radium-223 dichloride and atezolizumab from Cycle 2 onward.
  Interventions: Drug: Atezolizumab; Drug: Radium-223 Dichloride
- Cohort 2: ATZ + R-223-D (Staggered, 28-Day R-223-D Run-In) (Experimental): If Cohort 1 regimen is not tolerable, Arms A, B, and C will not be introduced and additional participants will be enrolled in this cohort to receive radium-223 dichloride in Cycle 1 and radium-223 dichloride and atezolizumab in Cycle 2. If the regimen is found to be safe, additional participants will be enrolled to receive this same treatment (radium-223 dichloride in Cycle 1 and radium-223 dichloride and atezolizumab from Cycle 2 onward). If, at Cycle 2, Cohort 2 regiment is not tolerable, additional participants will be enrolled in Cohort 3.
  Interventions: Drug: Atezolizumab; Drug: Radium-223 Dichloride
- Cohort 3: ATZ + R-223-D (Staggered, 56-Day R-223-D Run-In) (Experimental): If Cohort 2 regimen is not tolerable, additional participants will be enrolled in this cohort to receive radium-223 dichloride in Cycles 1, 2 and radium-223 dichloride and atezolizumab in Cycle 3. If the regimen is found to be safe, additional participants will be enrolled to receive this same treatment (radium-223 dichloride in Cycles 1, 2 and radium-223 dichloride and atezolizumab from Cycle 3 onward). If, at Cycle 3, Cohort 3 regiment is not tolerable, no additional participants will be enrolled in this study.
  Interventions: Drug: Atezolizumab; Drug: Radium-223 Dichloride

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be given at a dose of 840 milligrams (mg) via intravenous (IV) infusion on Days 1 and 15 of each 28-day cycle until loss of clinical benefit, unacceptable toxicity, or disease progression.
  Other Names: MPDL3280A
Drug: Radium-223 Dichloride — Radium-223 dichloride will be administered at a dose of 55 kilobecquerels per kilogram (kBq/kg) via slow IV bolus on Day 1 of each 28-day cycle for up to 6 cycles.
  Other Names: Xofigo

SUMMARY:
This study is designed to assess the safety and tolerability of atezolizumab when given in combination with radium-223 dichloride in participants with metastatic CRPC who have progressed after treatment with an androgen pathway inhibitor. This adaptive design study includes a cohort phase and a potential randomization phase. An initial concurrent dosing evaluation will evaluate the safety and tolerability of a treatment regimen that employs a concurrent start time for atezolizumab and radium-223 dichloride (Cohort 1). If concurrent dosing is found to be safe and tolerable in Cohort 1, additional participants will be enrolled and eligible participants will be randomized in a 1:1:1 ratio to Arms A, B, and C. If concurrent dosing is not tolerated in Cohort 1, new participants will be enrolled in a staggered dosing evaluation: Cohort 2 (28-day radium-223 dichloride run-in, atezolizumab will begin on Day 1 of Cycle 2) and Cohort 3 (56-day radium-223 dichloride run-in, atezolizumab will begin on Day 1 of Cycle 3). If the Cohort 2 schedule is tolerable, then additional participants will be enrolled using this treatment schedule; If the Cohort 2 schedule is not tolerable, subsequent participants will be enrolled in Cohort 3. If the Cohort 3 schedule is tolerable, then additional participants will be enrolled using this treatment schedule. If Cohort 3 schedule is not tolerable, no additional participant will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy greater than or equal to (>/=) 12 weeks
* Histologically confirmed, castrate-resistant adenocarcinoma of the prostate
* Measurable disease according to RECIST v1.1
* Multiple bone metastases within 12 weeks prior to study drug
* Participants receiving bisphosphonate or denosumab therapy must have been on a stable dose for at least 4 weeks
* Visceral metastasis and/or lymphadenopathy
* Tumors that are amenable to serial biopsy
* Disease progression according to Prostate Cancer Working Group 2 (PCWG2) criteria during or following treatment with at least one second generation androgen pathway inhibitor (for example, enzalutamide, abiraterone) for metastatic prostate cancer
* Adequate hematologic and end-organ function
* One prior taxane-containing regimen for mCRPC, or refusal or ineligibility of a taxane-containing regimen

Exclusion Criteria:

* History of small-cell or neuroendocrine prostate carcinoma
* Treatment with approved anti-cancer therapy (with the exception of abiraterone) within 3 weeks of study drug. Abiraterone must not be administered within 2 weeks prior to initiation of study treatment
* Participation in another clinical trial/investigation within 28 days prior to study drug
* Brain metastases or active leptomeningeal disease (with the exception of participants with treated epidural disease and no other epidural progression)
* Uncontrolled tumor-related pain
* Uncontrolled hypercalcemia
* Significant cardiovascular disease
* History of autoimmune disease except controlled/treated hypothyroidism, type 1 diabetes mellitus, or certain skin disorders
* Prior allogeneic stem cell or solid organ transplant
* History of pulmonary fibrosis/inflammation, including active tuberculosis
* Human immunodeficiency virus (HIV) or hepatitis B or C
* Prior treatment with cluster of differentiation (CD) 137 agonist, anti-programmed death (PD) 1, or anti-programmed death ligand (PD-L) 1 therapeutic antibody or pathway-targeting agents
* Immunostimulants within 4 weeks or immunosuppressants within 14 days prior to study drug
* Prior radium-223 dichloride or hemibody external radiotherapy
* Systemic strontium-89, samarium-153, rhenium-186, or rhenium-188 for bone metastases within 24 weeks prior to initiation of study treatment
* Spinal compression or structurally unstable bone lesions suggesting impending pathologic fractures based on clinical findings and/or magnetic resonance imaging (MRI)
* Bone marrow dysplasia
* Unmanageable fecal incontinence

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Dose-Limiting Toxicities (DLTs) | Days 1-28 of Cycle 1 (for Cohort 1), Cycle 2 (for Cohort 2), and Cycle 3 (for Cohort 3) (Cycle length = 28 days)
Percentage of Participants with Adverse Events (AEs) | From Screening to 90 days after the last dose (up to 42 months overall)
Percentage of Participants with Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | From Baseline until disease progression, death, loss to follow-up, withdrawal of consent, or study termination by the Sponsor, whichever occurs first (up to 42 months overall)

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of Atezolizumab | Pre-dose (0 hours) and 30 minutes post-dose (infusion length=60 minutes) on Day 1 of atezolizumab Cycle 1; pre-dose on Day 1 of atezolizumab Cycles 2, 3, 4, 8; at Treatment discontinuation and 120 days after last atezolizumab dose (up to 42 months)
Minimum Observed Serum Concentration (Cmin) of Atezolizumab | Pre-dose (0 hours) and 30 minutes post-dose (infusion length=60 minutes) on Day 1 of atezolizumab Cycle 1; pre-dose on Day 1 of atezolizumab Cycles 2, 3, 4, 8; at Treatment discontinuation and 120 days after last atezolizumab dose (up to 42 months)
Percentage of Participants with Anti-Therapeutic Antibodies (ATAs) to Atezolizumab | Pre-dose (0 hours) on Day 1 of atezolizumab Cycles 1, 2, 3, 4, 8; at treatment discontinuation (up to 36 months); and 120 days after last atezolizumab dose (up to 42 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- United States (17):
  - City of Hope, Duarte, California
  - University of California, San Francisco, Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Yale School of Medicine, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic Hospital - Florida, Jacksonville, Florida
  - Indiana University Health Melvin & Bren Simon Cancer Center, Indianapolis, Indiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic - Minnesota, Rochester, Minnesota
  - Comprehensive Cancer Centers of Nevada (CCCN) - Central Valley, Las Vegas, Nevada
  - Memorial Sloan-Kettering Cancer Center, Commack, New York
  - Duke University Hospital, Durham, North Carolina
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Fong L, Morris MJ, Sartor O, Higano CS, Pagliaro L, Alva A, Appleman LJ, Tan W, Vaishampayan U, Porcu R, Tayama D, Kadel EE 3rd, Yuen KC, Datye A, Armstrong AJ, Petrylak DP. A Phase Ib Study of Atezolizumab with Radium-223 Dichloride in Men with Metastatic Castration-Resistant Prostate Cancer. Clin Cancer Res. 2021 Sep 1;27(17):4746-4756. doi: 10.1158/1078-0432.CCR-21-0063. Epub 2021 Jun 9. PMID 34108181